CLINICAL TRIAL: NCT00442117
Title: A Comparison of Mometasone Furoate DPI Versus Budesonide DPI in Mild Persistent and Moderate Persistent Asthmatic Patients
Brief Title: A Comparison of Mometasone Furoate DPI Versus Budesonide DPI in Budesonide DPI in Asthmatics (Study P04880)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P04880
Record Dates: First submitted 2007-02-28; First posted 2007-03-01 (Estimated); Results first posted 2011-02-10 (Estimated); Last update posted 2024-05-20 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma | interventions — Mometasone Furoate; Budesonide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MF-DPI (Experimental): MF DPI 200 mcg, two puffs once daily PM (total of 400 mcg/day)
  Interventions: Drug: mometasone furoate dry powder inhaler
- BUD-DPI (Active Comparator): Budesonide (BUD) DPI 200 mcg, two puffs twice daily (total of 800 mcg/day)
  Interventions: Drug: Budesonide DPI

INTERVENTIONS:
Drug: mometasone furoate dry powder inhaler — MF DPI 200 mcg, two puffs once daily PM (total of 400 mcg/day) for 12 weeks.
  Other Names: Asmanex
  Arms: MF-DPI
Drug: Budesonide DPI — Budesonide (BUD) DPI 200 mcg, two puffs twice daily (total of 800 mcg/day) for 12 weeks.
  Other Names: Pulmicort
  Arms: BUD-DPI

SUMMARY:
This study will be an open-label, parallel-group comparison of Mometasone Furoate Dry Powder Inhaler (MF-DPI) 200 mcg once daily in the evening with two puffs vs. Budesonide Dry Powder Inhaler (BUD-DPI) 200 mcg twice daily with two puffs each time in patients previously treated with inhaled corticosteroids (ICS) or without ICS with diagnosed mild persistent or moderate persistent asthma (classified as Global Initiative For Asthma, 2005) in the previous 4 weeks. The primary efficacy endpoint is percent change from baseline in FEV1.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 12 years of age or older of either gender, who (and their parent/guardian if the subject is under the age of 20) must demonstrate their willingness to sign and write informed consent.
* Subjects must have had a history of asthma for at least 6 months.
* The subject must be diagnosed mild persistent or moderate persistent asthma and his/her FEV1 must be >= 60% of predicted normal at both the Screening and Baseline visits, when short-acting inhaled beta agonists have been withheld for at least six hours and long-acting inhaled beta agonists have been withheld for at least 12 hours.
* Subjects must demonstrate an increase in absolute FEV1 of >= 12%, with an absolute volume increase of at least 200 mL, after reversibility testing at the Screening visit, or historically within the past 12 months; Subjects without documented absolute FEV1 of >= 12% in reversibility test within the past 12 months need to demonstrate a positive result in Methacholine challenge test.
* If Subjects with ICS treatment have been using ICS on a daily basis for at least 4 weeks prior to Screening. For the two weeks prior to Screening, subjects must have been on a stable regimen of ICS. Each ICS dose is shown in following:

  * Flunisolide between 1000 to 2000 mcg/day
  * Budesonide between 400 to 800 mcg/day
  * Triamcinolone acetonide between 600 to 1600 mcg/day
  * Beclomethasone Dipropionate between 252 to 840 mcg/day
  * Fluticasone propionate between 200 to 500 mcg/day
* Women of childbearing potential must have a negative urine (hCG) pregnancy test on the day of randomization (Baseline visit).
* Women of childbearing potential (includes women who are less than 1 year postmenopausal) must be using or agree to use an acceptable method of birth control (e.g., hormonal contraceptive, medically prescribed IUD, condom in combination with spermicide) or be surgically sterilized (e.g., hysterectomy or tubal ligation) if they become sexually active.
* Subjects must understand and be able to adhere to visit schedules and enter information in a daily diary.

Exclusion Criteria:

* Female subjects who are pregnant, breast-feeding, or are pre-menarcheal.
* Subjects who are heavy smokers (more than 10 pack years) or who smoked within previous 6 months.
* Subjects who have required daily or alternate day oral corticosteroid treatment for more than a total of 14 days during the 3 months immediately prior to the Screening visit, and/or subjects who have required a course of systemic corticosteroids within the previous month.
* Subjects who used Leukotriene modifiers within 2 weeks of screening.
* Subjects who took immunosuppressive agents within the previous 3 months.
* Subjects who use daily nebulized ß2-adrenergic agonists.
* Subjects who have had either an asthma exacerbation or a clinically relevant change in asthma medication within the last 4 weeks.
* Subjects who have been admitted to the hospital for asthma control within the previous 3 months or have needed emergency service for asthma more than once within the previous 6 months.
* Subjects who have required ventilator support for respiratory failure secondary to their asthma within the last 5 years.
* Subjects who have used any investigational drug in the 30 days prior to Baseline, or subjects who have been treated with any investigational antibody for asthma in the 90 days prior to Baseline.
* Subjects who are allergic or have had an idiosyncratic reaction to corticosteroids.
* Subjects with evidence of clinically significant oropharyngeal candidiasis at Screening or Baseline.
* Subjects with any clinically significant disorder of the cardiovascular, neurologic, hematologic, gastrointestinal, cerebrovascular, or immunologic system, or respiratory disease other than asthma (e.g. COPD), or any other disorder which may interfere with the study evaluations or affect subject safety.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 180 (Actual)
Dates: Start 2007-06; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 180 participants were enrolled and randomized. There were 8 participants who had taken at least one dose of study medication, but were not eligible for the study and therefore were withdrawn, resulting in the Intent-to-Treat (ITT) population of 172 participants.
Groups:
- MF-DPI: Mometasone Furoate Dry Powder Inhaler (MF DPI) 200 mcg, two puffs once daily in the evening (PM) (total of 400 mcg/day)
- BUD-DPI: Budesonide Dry Powder Inhaler (BUD DPI) 200 mcg, two puffs twice daily (total of 800 mcg/day)
Period: Overall Study
Arm/Group | MF-DPI | BUD-DPI
Started | 85 | 87
Completed | 47 | 49
Not Completed | 38 | 38
Not completed — Adverse Event | 3 | 2
Not completed — Lack of Efficacy | 2 | 6
Not completed — Lost to Follow-up | 1 | 2
Not completed — Withdrawal by Subject | 2 | 2
Not completed — Major Deviation | 25 | 20
Not completed — Non compliance with protocol | 3 | 5
Not completed — Met Withdrawal Criteria | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MF-DPI | BUD-DPI | Total
Number analyzed (Participants) | 91 | 89 | 180
Age, Customized [Number; unit: participants] — Number of participants analyzed includes data of the total enrolled population
  participants | 91 | 89 | 180
Sex: Female, Male [Count of Participants; unit: Participants] — Number of participants analyzed includes data of the total enrolled population
  Participants
    Female | 48 | 40 | 88
    Male | 43 | 49 | 92

OUTCOME MEASURES:

1. Primary Outcome: Mean Percent Change of Forced Expiratory Volume in One Second (FEV1) From Baseline to Week 12.
Description: FEV1 (forced expiratory volume in one second) measurement at the Baseline visit was compared to the FEV1 measurement during the last visit at Week 12. The mean percent change was calculated.
Time Frame: Baseline and Week 12
Population: Intent-to treat (ITT) population: All randomized patients who have taken at least one dose of study medication and have at least one post-baseline efficacy information.
Measure: Mean (Standard Deviation); unit: Percent Change of FEV1
Arm/Group | MF-DPI | BUD-DPI
Number analyzed (Participants) | 85 | 87
Percent Change of FEV1 | -1.09 (10.57) | -0.02 (10.17)
Statistical Analysis 1: Comparison: MF-DPI vs BUD-DPI; Test type: Superiority or Other; p = 0.4982, ANOVA; Mean Difference (Final Values) = -1.074, 95% CI 2-sided [-4.196 to 2.049]

2. Secondary Outcome: Mean Percent Change of FVC (Forced Vital Capacity) From Baseline to Week 12.
Description: The FVC measurement at the baseline was compared to the FVC measurement during the last visit at Week 12. The mean percent change was calculated.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change of FVC
Arm/Group | MF-DPI | BUD-DPI
Number analyzed (Participants) | 85 | 87
Percent Change of FVC | -0.11 (10.91) | -0.88 (11.50)
Statistical Analysis 1: Comparison: MF-DPI vs BUD-DPI; Test type: Superiority or Other; p = 0.6544, ANOVA; Mean Difference (Final Values) = 0.7601, 95% CI 2-sided [-2.585 to 4.106]

3. Secondary Outcome: Mean Percent Change of Forced Expiratory Flow (FEF) at (25-75% Interval) From Baseline to Week 12.
Description: The FEF (25-75%) measurement at the baseline was compared to the FEF (25-75%) measurement during the last visit at Week 12. The mean percent change was calculated.
Time Frame: Baseline and Week 12
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent Change of FEF
Arm/Group | MF-DPI | BUD-DPI
Number analyzed (Participants) | 85 | 87
Percent Change of FEF | 0.01 (12.68) | 1.72 (12.92)
Statistical Analysis 1: Comparison: MF-DPI vs BUD-DPI; Test type: Superiority or Other; p = 0.3796, ANOVA; Mean Difference (Final Values) = -1.704, 95% CI 2-sided [-5.528 to 2.115]

4. Secondary Outcome: Mean Percent Change of AM PEFR (Peak Exploratory Flow Rate) From Baseline to Week 12.
Description: The AM PEFR measurement at the Baseline visit was compared to the AM PEFR measurement during the last visit at Week 12. The mean percent change was calculated.
Time Frame: Baseline and Week 12
Population: Intent-to treat (ITT) population: All randomized patients who have taken at least one dose of study medication and have at least one post-baseline efficacy information. Two participants in the MF-DPI group and three participants in the BUD-DPI group were excluded from the analysis.
Measure: Mean (Standard Deviation); unit: Percent Change of AM PEFR
Arm/Group | MF-DPI | BUD-DPI
Number analyzed (Participants) | 83 | 84
Percent Change of AM PEFR | 2.59 (42.36) | 1.93 (71.02)
Statistical Analysis 1: Comparison: MF-DPI vs BUD-DPI; Test type: Superiority or Other; p = 0.9622, ANOVA; Mean Difference (Final Values) = 0.432, 95% CI 2-sided [-17.560 to 18.240]

ADVERSE EVENTS:
Arm/Group | MF-DPI | BUD-DPI
Serious Adverse Events (participants affected / at risk) | 3/91 | 2/89
Other Adverse Events (participants affected / at risk) | 13/91 | 15/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF-DPI (N=91) | BUD-DPI (N=89)
cellulitis (Infections and infestations) | 2 (2) | 0 (0)
pregnancy test positive (Investigations) | 0 (0) | 1 (1)
spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
nasal polyps (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MF-DPI (N=91) | BUD-DPI (N=89)
upper respiratory tract infection (Infections and infestations) | 13 (14) | 15 (15)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No